CLINICAL TRIAL: NCT00208364
Title: Uncontrolled Prospective Multi-Centre Post Marketing Surveillance Study to Monitor the Long Term Survivorship of Pinnacle Acetabular Cup Prosthesis With a Metal on Metal Bearing in Subjects With Aetiologies Requiring a Primary Total Hip Replacement
Brief Title: A Two Centre Study to Assess the Long-term Performance of the Pinnacle™ Cup With a Metal-on-Metal Bearing in Primary Total Hip Replacement
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated early due to business reasons
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT01/11
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Post-traumatic Arthritis; Collagen Disorders; Avascular Necrosis; Traumatic Femoral Fractures; Nonunion of Femoral Fractures; Congenital Hip Dysplasia; Slipped Capital Femoral Epiphysis
Keywords: Hip; Cementless; Metal-on-Metal
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Collagen Diseases; Osteonecrosis; Hip Dislocation, Congenital; Slipped Capital Femoral Epiphyses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pinnacle Acetabular Cup System (Other): A cementless acetabular cup with metal liner for use in total hip replacement
  Interventions: Device: Pinnacle Acetabular Cup System

INTERVENTIONS:
Device: Pinnacle Acetabular Cup System — A cementless acetabular cup with metal liner for use in total hip replacement

SUMMARY:
The purpose of this study is to monitor the performance and determine the metal ion release of the Pinnacle™ Cup with a metal-on-metal bearing combination in the treatment of patients with hip joint disease requiring a total hip replacement. Patients who enter the study will be evaluated at regular intervals following hip surgery using patient, clinical and x-ray assessments. A subset of patients will also have blood samples taken at regular intervals to allow the metal ion levels to be determined.

ELIGIBILITY:
Inclusion Criteria:

i) Male or female subjects, aged between 18 and 70 years inclusive.

ii) Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.

iii) Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.

iv) Subjects undergoing primary total hip replacement who are suitable for cementless acetabular components.

Exclusion Criteria:

i) Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.

ii) Subjects undergoing revision hip replacement.

iii) Women who are pregnant.

iv) Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.

v) Subjects who have participated in a clinical study with an investigational product in the last 12 months.

vi) Subjects who are currently involved in any injury litigation claims.

Additional Exclusion Criteria for Subjects Having Blood Analysis:

1. Subjects who currently have other metallic foreign bodies including trauma products and joint arthroplasties unless known to be pure titanium or titanium alloy.
2. Subjects with an occupational exposure to cobalt or chromium.
3. Subjects who have ingested medication or vitamins containing cobalt or chromium within the last 12 months.
4. Subjects who, in the opinion of the Investigator, will possibly require a separate joint replacement operation within the next two years, including revision operations.
5. Subjects who are undergoing a simultaneous bilateral total hip replacement.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2004-04; Primary Completion 2014-10 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Kaplan-Meier survivorship calculated at the 5 year time point. | 5 years

SECONDARY OUTCOMES:
Annual Kaplan-Meier survivorship calculationsMetal ion analysis in whole blood | Annually
Harris Hip score | 6mths, 1yr, 2yrs, 3yrs, 5yrs, 7yrs 10yrs and 15yrs post-surgery
Oxford Hip score | 6mths, 1yr, 2yrs, 3yrs, 5yrs, 7yrs 10yrs and 15yrs post-surgery
Radiological analysis | 6mths, 1yr, 2yrs, 3yrs, 5yrs, 7yrs 10yrs and 15yrs post-surgery
Metal ion analysis in whole blood | pre-discharge, 6mths, 1yr, 2 yrs and 5yrs post-surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Ospedale Riuniti Di Bergamo, Bergamo, Italy
- Royal Orthopaedic Hospital, Birmingham, United Kingdom